CLINICAL TRIAL: NCT00921778
Title: Long-Term Outcome Following Laparoscopic Supracervical Hysterectomy Performed With and Without Excision of the Endocervix in a Reverse Cone Pattern
Acronym: LSH-LAPCONE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ullevaal University Hospital (Other)
Responsible Party: Ullevaal University Hospital, Oslo University Hostpital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LSH-LAPCONE UUS
Record Dates: First submitted 2009-06-15; First posted 2009-06-16 (Estimated); Last update posted 2009-06-16 (Estimated); Status verified 2008-08

CONDITIONS: Vaginal Bleeding
Keywords: Laparoscopic supracervical hysterectomy; Vaginal bleeding; Patient satisfaction; vaginal bleeding after laparoscopic hysterectomy
MeSH Terms: conditions — Uterine Hemorrhage; Patient Satisfaction

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Lapcone — Use of Lapcone during LSH
Procedure: laparoscopic supracervical hysterectomy — laparoscopic supracervical hysterectomy

SUMMARY:
The occurrence of persistent vaginal bleeding following laparoscopic supracervical hysterectomy (LSH) is reported in the wide range of 0 % - 25 %. Experienced gynaecologists have claimed that removal of any remaining endometrium in a reverse cone pattern at the time of the hysterectomy reduces the occurrence of persistent vaginal bleeding to a minimum. The effect of this particular technique has not been reported.

Ullevaal University Hospital have developed an unipolar electrode for this study (Lapcone electrode, mod. UUS, L: 25cm, 6x10, Art. No. REM-270, Ross Electro Medical Ltd, Unit K1&K2, Quarry Fields Estate, Mere, Wiltshire BA12 6LA, London, UK). The electrode is CE approved.

Outcome: 1.Occurrence of vaginal bleeding 12 months after the procedure. 2. Patient satisfaction 12 months after the procedure (10-point analogue scale).

Design: Prospective randomised trial. Methods; The study participants are randomised to laparoscopic supracervical hysterectomy performed by perioperative electrocoagulation from the upper cervical canal (n=70) or performed by excision of the endocervix in a reverse cone pattern followed by electrocoagulation of the upper cervical canal (n =70).

ELIGIBILITY:
Inclusion Criteria:

* All premenopausal women who are referred to the departement due to a benign condition requiring hysterectomy and who have given informed consent are eligible for study recruitment

Exclusion Criteria:

* Women who are unable to communicate in written Norwegian or oral English language.
* Woman with a previous history of cervical dysplasia, with cellular changes suggestive of dysplasia in preoperative smear or wtih atypical hyperplasia og malignancy in preoperative endometrial biopsy
* Women who after a thorough clinical evaluation are found to be more suited for vaginal, abdominal or total hysterectomy
* Women with a coexisting condition requiring no remaining ovaries after the procedure
* Postmenopausal women
* Women using hormone therapy (HT)

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2008-09; Primary Completion 2010-12 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Occurrence of vaginal bleeding 12 months after the procedure. | 12 months after operation

SECONDARY OUTCOMES:
Patient satisfaction 12 months after the procedure (10-point analogue scale). | 12 months after operation

CONTACTS AND LOCATIONS:
Locations (1):
- Ullevaal University Hospital, Oslo, Norway

REFERENCES:
- See also: homepage Ullevaal University Hospital — http://www.ulleval.no